CLINICAL TRIAL: NCT01237912
Title: A European, Multi-centre Study to Determine the Exposure of Adult Smokers and Non-smokers to Cigarette Smoke Constituents
Brief Title: European Exposure Study
Status: Completed | Type: Observational
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: SPA0403
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The current study was designed to determine the exposure of adult smokers and non-smokers to cigarette smoke constituents through evaluation of selected biomarkers of exposure.

DETAILED DESCRIPTION:
The purpose of the study was to provide a greater knowledge about human exposure to cigarette smoke constituents by evaluating selected biomarkers of exposure in smokers and non-smokers. This was an observational, parallel-group study to be conducted at multiple centres in the UK, Germany, and Switzerland. It was planned to enrol sufficient subjects such that at least 1440 subjects complete the study.

ELIGIBILITY:
Inclusion Criteria:

Smokers: Subjects who smoked commercial cigarettes exclusively (less than or equal to 10 mg ISO tar yield in Germany and the UK; less than or equal to 12 mg ISO tar yield in Switzerland) with a regular consumption of at least 1 cigarette per day over the last 12 months without change in brand over the previous 3 months.

or

Non-smokers: Subjects who did not smoke commercial cigarettes, hand-rolled cigarettes, cigars, pipes, bidis, and did not use other nicotine-containing products (patch, gum, lozenges etc.) within 1 year prior to Visit 1 and throughout the study duration.

Exclusion Criteria:

* Female subjects with child-bearing potential were to be excluded if

  1. Subject was pregnant (or did not have negative pregnancy tests) or breast-feeding
  2. Subject did not agree to use an acceptable method of contraception

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female 21 years of age or older with a stable health status as determined by the Investigator and who were able to understand the subject information and to comply with the study procedures and study schedule.
Sampling Method: Non-Probability Sample
Enrollment: 1667 (Actual)
Dates: Start 2005-04; Primary Completion 2006-05 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine the exposure of adult smokers and non-smokers to cigarette smoke constituents | 2 consecutive visits within 14 days
  To determine the exposure of adult smokers and non-smokers to the following cigarette smoke constituents: carbon monoxide, nicotine, acrolein, benzene, 1,3-butadiene, 4-aminobiphenyl (4-ABP), 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK), o-toluidine, pyrene (1-OHP), 2-aminonaphthalene (2-NA).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Smith, Principal Investigator — Celerion, 22-24 Lisburn Road, Belfast, BT9 6AD, Northern Ireland
Locations (1):
- Stephen Smith, Belfast, Northern Ireland, United Kingdom

REFERENCES:
- [Result] Lindner D, Smith S, Leroy CM, Tricker AR. Comparison of exposure to selected cigarette smoke constituents in adult smokers and nonsmokers in a European, multicenter, observational study. Cancer Epidemiol Biomarkers Prev. 2011 Jul;20(7):1524-36. doi: 10.1158/1055-9965.EPI-10-1186. Epub 2011 May 25. PMID 21613391